CLINICAL TRIAL: NCT05902962
Title: A Phase 1 Open-Label, Single Arm Dose Escalation Study to Evaluate the Safety and Tolerability of Intravitreally Administered VP-001 in Participants With Confirmed PRPF31 Mutation-Associated Retinal Dystrophy
Brief Title: SAD of IVT VP-001 in PRPF31 Mutation-Associated Retinal Dystrophy Subjects
Acronym: Platypus
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP001-CL101
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Retinal Dystrophy; PRPF31 Mutationassociated Retinal Dystrophy; RP11
MeSH Terms: conditions — Retinal Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm dose escalation study of VP-001 (Experimental)
  Interventions: Drug: VP-001

INTERVENTIONS:
Drug: VP-001 — Phase 1 open-label, single arm dose escalation study of VP-001 in participants with genetically confirmed PRPF31 mutation-associated retinal dystrophy

SUMMARY:
A Phase 1 Open-Label, Single Arm Dose Escalation Study to Evaluate the Safety and Tolerability of Intravitreally Administered VP-001 in Participants with Confirmed PRPF31 Mutation-Associated Retinal Dystrophy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female sex; ≥ 18 years of age at Baseline (Visit 2).
2. Have a molecular (genetic) diagnosis of PRPF31 mutation.
3. Have a clinical diagnosis of PRPF31 mutation-associated retinal dystrophy, that is, RP11. The following conditions are allowed for inclusion if due to RP11, if in the opinion of the investigator they will not interfere with study evaluations or have resolved: macular edema (intraretinal, sub-retinal or other fluid) requiring regular treatment at a frequency of less than every 6 weeks; macular edema must be stable for at least 3 months prior to Screening (Visit 1). The investigator must consult with the study Medical Monitor.
4. If ≥ 18 years of age, understand the language of the informed consent and are willing and able to provide written informed consent prior to any study procedures. Are willing to comply with the instructions and attend all scheduled study visits.

6. Have light perception (LP) or better vision in the study eye. 7. Participants of childbearing potential and male participants must not be pregnant or lactating and must be sexually inactive by abstinence, which is consistent with the preferred and usual lifestyle of the participant or agree to use adequate birth control throughout study duration. Adequate birth control is defined as hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a condom or diaphragm; intrauterine device (IUD); or surgical sterilization of partner. For nonsexually active participants, abstinence may be regarded as an adequate method of birth control. Participants of childbearing potential include all participants who have experienced menarche and have not undergone successful surgical sterilization (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) or are not post-menopausal (12 months after last menses).

Exclusion Criteria:

1. Have any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study that include but are not limited to infection, uncontrolled elevated blood pressure, cardiovascular disease, or glycemic control issues, or any other medical condition that may put the participant at risk due to study procedures.
2. Mutations in genes that cause autosomal dominant RP, X-linked RP, or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than PRPF31 mutations.
3. Have used anti-vascular endothelial growth factor (VEGF) agents within 2 months or corticosteroid injections within the last 3 months.
4. Have had Ozurdex® implants placed within 3 months or Retisert® or Iluvien® implants placed within 3 years prior to Baseline (Visit 2).
5. Within 3 months prior to Baseline (Visit 2), have undergone any vitreoretinal surgery (scleral buckle, pars plana vitrectomy, retrieval of a dropped nucleus or intraocular lens, radial optic neurotomy, sheathotomy, cyclodestructive procedures or multiple filtration surgeries [2 or more]) or any other ocular surgery.
6. Have ocular media opacity or poor pupillary dilation prohibiting quality ophthalmic evaluation or photography, as assessed by the investigator.
7. Have used any investigational drug or device within 90 days or 5 estimated half-lives of Baseline (Visit 2), whichever is longer, or plan to participate in another study of drug or device during the study period. Participation in observational trials is allowable based on investigator discretion and consultation with the Medical Monitor. It is assumed that the observational trial evaluations would not interfere with participation in this study.
8. Have received any prior cell or gene therapy for a retinal condition.
9. Have a recent history (<6 months) or current excessive recreational drug or alcohol use, in the opinion of the investigator.
10. Any retinal pathology other than RP11 that in the investigator's opinion could affect study results.
11. Participants should not have any conditions, in the investigator's opinion, that may put the participant at increased risk, confound study data, or interfere significantly with the participant's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The incidence, severity, and relatedness of treatment-emergent ocular adverse events (TEAEs) and treatment-emergent serious adverse events (TE-SAEs) in the study eye | over a 24-week time period
The incidence, severity, and relatedness of treatment-emergent ocular adverse events (TEAEs) and treatment-emergent serious adverse events (TE-SAEs) in the study eye | over a 48-week time period

SECONDARY OUTCOMES:
Adverse Events and Treatment Emergent Serious adverse events (SAEs) in the fellow eye | over a 24-week time period
Adverse Events and Treatment Emergent serious adverse events (SAEs) in the fellow eye | over a 48-week time period
Incidence, severity relatedness and of non-ocular TEAEs | over a 24-week time period
Incidence, severity relatedness and of non-ocular TEAEs | over a 48-week time period

OTHER OUTCOMES:
Change from Baseline in Best-corrected visual acuity (BCVA) letter score using Early Treatment Diabetic Retinopathy Study (ETDRS) charts | over a 24-week time period
Change from Baseline in Best-corrected visual acuity (BCVA) letter score using Early Treatment Diabetic Retinopathy Study (ETDRS) charts | over a 48-week time period
Change from Baseline in lowest passing light level using Ora-VNC™ mobility test | over a 24-week time period
Change from Baseline in lowest passing light level using Ora-VNC™ mobility test | over a 48-week time period
Change from Baseline in Low luminance visual acuity (LLVA) letter score | over a 24-week time period
Change from Baseline in Low luminance visual acuity (LLVA) letter score | over a 48-week time period
Change from Baseline in Visual field sensitivity as measured by static perimetry with topographic analysis (Hill of Vision) | over a 24-week time period
Change from Baseline in Visual field sensitivity as measured by static perimetry with topographic analysis (Hill of Vision) | over a 48-week time period
Change from Baseline in Mean retinal sensitivity as measured by fundus-guided microperimetry | over a 24-week time period
Change from Baseline in Mean retinal sensitivity as measured by fundus-guided microperimetry | over a 48-week time period
Change from Baseline in Visual fields as measured by kinetic perimetry, utilizing I4e, III4e and V4e stimuli | over a 24-week time period
Change from Baseline in Visual fields as measured by kinetic perimetry, utilizing I4e, III4e and V4e stimuli | over a 48-week time period
Change from Baseline in Rod- and cone-mediated retinal function as measured by white, red and blue FST | over a 24-week time period
Change from Baseline in Rod- and cone-mediated retinal function as measured by white, red and blue FST | over a 48-week time period
Change from Baseline in Retinal thickness on SD-OCT, including retinal thickness in each ETDRS subfield and ellipsoid zone (EZ) area and volume | over a 24-week time period
Change from Baseline in Retinal thickness on SD-OCT, including retinal thickness in each ETDRS subfield and ellipsoid zone (EZ) area and volume | over a 48-week time period
Change from Baseline in Participant reported outcome measures utilizing the Patient Global Impressions of Change (PGI-C) and Patient Global Impressions of Severity (PGI-S) | over a 24-week time period
Change from Baseline in Participant reported outcome measures utilizing the Patient Global Impressions of Change (PGI-C) and Patient Global Impressions of Severity (PGI-S) | over a 48-week time period
Change from Baseline in Retinal function using full-field electroretinography (ERG) | over a 24-week time period
Change from Baseline in Retinal function using full-field electroretinography (ERG) | over a 48-week time period
Change from Baseline in Area of hypo-autofluorescence captured by FAF | over a 24-week time period
Change from Baseline in Area of hypo-autofluorescence captured by FAF | over a 48-week time period
Change from Baseline in Abnormalities captured by wide-field fundus photography | over a 24-week time period
Change from Baseline in Abnormalities captured by wide-field fundus photography | over a 48-week time period

CONTACTS AND LOCATIONS:
Overall Officials: Sreenivasu Mudumba, Study Chair — PYC
Locations (6):
- United States (6):
  - University of Florida Health, Jacksonville, Florida
  - Bascom Palmer Eye Institute University of Miami, Miami, Florida
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Oregon Health and Science University - Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine- Alkek Eye Center, Houston, Texas